CLINICAL TRIAL: NCT00004874
Title: Expanded Access Study of Iodine-131 Anti-B1 Antibody for Relapsed/Refractory Low-Grade and Transformed Low-Grade Non-Hodgkin's Lymphoma
Brief Title: Monoclonal Antibody Therapy in Treating Patients With Non-Hodgkin's Lymphoma
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: lack of FDA approval
Sponsor: University of Nebraska (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Coulter Pharmaceutical, Inc. (Industry)
Responsible Party: Principal Investigator, Julie M Vose, MD, Principal Investigator, University of Nebraska
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 259-98; P30CA036727 (NIH); UNMC-259-98; COULTER-CP-98-020
Record Dates: First submitted 2000-03-07; First posted 2003-12-16 (Estimated); Last update posted 2018-01-17 (Actual); Status verified 2018-01

CONDITIONS: Lymphoma
Keywords: recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent small lymphocytic lymphoma
MeSH Terms: conditions — Lymphoma; Lymphoma, Follicular; Leukemia, Lymphocytic, Chronic, B-Cell | interventions — tositumomab I-131

INTERVENTIONS:
Radiation: tositumomab and iodine I 131 tositumomab — Dosimetric Dose:Unlabeled anti-B1 (450mg) will be given as peripheral or central IV infusion over one hour or longer depending upon rate-dependent side effects. A trace-labeled dose of 131I-anti-B will be infused over 20 minutes, if rate-dependent side effects permit. An amount of unlabeled Anti-B1 Antibody is added to the 5 mCi of Iodine-131 Anti-B1 Antibody sufficient to result in a final amount of 35 mg of Anti-B1 antibody. On study Day 7 (may be delayed up to study Day 14), patients will receive the therapeutic dose, which consists of an infusion of 450mg of Anti-B1 Antibody followed by an infusion of Iodine-131 Anti-B1 Antibody.
  Other Names: Iodine-131 Anti-B1 Antibody

SUMMARY:
RATIONALE: Monoclonal antibodies can locate cancer cells and either kill them or deliver cancer-killing substances to them without harming normal cells.

PURPOSE: Phase III trial to determine the effectiveness of monoclonal antibody therapy in treating patients who have relapsed or refractory non-Hodgkin's lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the efficacy and safety of iodine I 131 monoclonal antibody anti-B1 in patients with relapsed or refractory, low grade or transformed low grade B-cell non-Hodgkin's lymphoma.

OUTLINE: On day 1, patients receive unlabeled monoclonal antibody anti-B1 (MOAB anti-B1) IV over 1 hour followed by a tracer dose of iodine I 131 MOAB anti-B1 IV over 30 minutes to determine biodistribution and a therapeutic dose of iodine I 131 MOAB anti-B1. Patients receive unlabeled MOAB anti-B1 IV over 1 hour followed by a therapeutic dose of iodine I 131 MOAB anti-B1 IV over 30 minutes on day 8. Patients are followed at weeks 13 and 25 and then every 6 months for up to 2 years.

PROJECTED ACCRUAL: Expanded Access Trial, no maximum accrual

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically proven relapsed or refractory, low grade or transformed low grade B-cell non-Hodgkin's lymphoma including the following: Small lymphocytic Follicular small cleaved cell Follicular mixed small cleaved and large cell (less than 50% large cell component) Tumor must be positive for CD20 antigen Relapse or disease progression following at least 1 chemotherapy regimen or failure to achieve an objective response (complete or partial response) on prior chemotherapy regimen No disease progression, within 1 year of irradiation, arising in a field previously irradiated with more than 3500 cGy Mean of no greater than 25% intratrabecular marrow space involved with lymphoma on bilateral iliac crest bone marrow biopsy A new classification scheme for adult non-Hodgkin's lymphoma has been adopted by PDQ. The terminology of "indolent" or "aggressive" lymphoma will replace the former terminology of "low", "intermediate", or "high" grade lymphoma. However, this protocol uses the former terminology.

PATIENT CHARACTERISTICS: Age: 19 and over Performance status: Karnofsky 60-100% Life expectancy: At least 3 months Hematopoietic: Absolute neutrophil count at least 1,500/mm3 Platelet count at least 100,000/mm3 Hepatic: Bilirubin less than 1.5 times upper limit of normal (ULN) AST less than 5 times ULN Renal: Creatinine less than 1.5 times ULN No active obstructive hydronephrosis Cardiovascular: No New York Heart Association class III or IV heart disease Other: No active infection requiring IV antibiotics No other concurrent illness that would preclude evaluation No prior malignancy within the past 5 years except adequately treated skin cancer, carcinoma in situ of the cervix, or lymphoma HIV negative Not pregnant or nursing Negative pregnancy test Fertile patients must use effective contraception during and for 6 months after study No prior allergic reaction to iodine other than IV iodine containing contrast materials Human antimouse antibody negative

PRIOR CONCURRENT THERAPY: Biologic therapy: At least 4 weeks since prior immunotherapy or cytokine treatment and recovered No prior hematologic stem cell transplantation Chemotherapy: See Disease Characteristics At least 4 weeks since prior chemotherapy (at least 6 weeks since prior nitrosoureas) and recovered Endocrine therapy: Not specified Radiotherapy: See Disease Characteristics At least 4 weeks since prior radiotherapy and recovered No prior radioimmunotherapy Surgery: Not specified Other: No concurrent IV antibiotics

Ages: 19 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 1998-11; Primary Completion 2002-04 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Expanded Access | Study completion
  The primary objective of this stud is to make Iodin-131 Anti-B1 Antibody more broadly available to patients

SECONDARY OUTCOMES:
Safety | Study completion
  Secondary endpoints of the study will be to obtain additional information on the safety of Iodine-131 Anti-B1 Antibody
efficacy | study completion
  Secondary endpoints of the study will be to obtain additional information on the efficacy of Iodine-131 Anti-B1 Antibody

CONTACTS AND LOCATIONS:
Overall Officials: Julie M. Vose, MD, Study Chair — University of Nebraska
Locations (1):
- University of Nebraska Medical Center, Omaha, Nebraska, United States